CLINICAL TRIAL: NCT04567966
Title: Cortical Bone Plate Versus Cortico-cancellous Block Graft for Horizontal Ridge Augmentation: Histomorphometric and Cone Beam Computed Tomography Study
Brief Title: Cortical Bone Plate Versus Cortico-cancellous Block Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mina Adel Rizk Botros, Assistant Researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER 18-1D
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Horizontal Atrophy of Edentulous Alveolar Ridge
Keywords: Split-bone block technique; Cortical bone plate; Cortico-cancellous block graft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cortical bone plate (Experimental): A cortical plate was harvested from the external oblique ridge and split in half. Then one plate was fixed at a distance from the atrophied ridge and autogenous bone chips were used to fill the gap between the plate and the ridge.
  Interventions: Procedure: Split-block technique
- Cortico-cancellous block graft (Active Comparator): A cortico-cancellous block graft was harvested from the symphysis of the mandible and fixed to the atrophied ridge.
  Interventions: Procedure: Cortico-cancellous block graft

INTERVENTIONS:
Procedure: Split-block technique — Horizontal ridge augmentation using the split-block technique where a cortical bone plate harvested from the external oblique ridge was split in half and fixed at a distance from the atrophied ridge. Then autogenous bone chips were packed in the gap between the plate and the ridge.
  Arms: Cortical bone plate
Procedure: Cortico-cancellous block graft — Horizontal ridge augmentation using a cortico-cancellous block harvested from the chin of the mandible.
  Arms: Cortico-cancellous block graft

SUMMARY:
Horizontal ridge augmentation using either cortical bone plate technique or cortico-cancellous block graft was the aim of the study. Bone quality was analyzed histomorphomterically, and horizontal dimensional changes were assessed using CBCT.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients aged 18 years or older with partial edentulism of the mandible
* The residual ridge width must be 4 mm or less
* Intra-oral donor sites should be available in the external oblique ridge and symphyseal area

Exclusion Criteria:

* Patients with general contraindications for implant surgery such as uncontrolled diabetes
* Irradiation of the head and neck region
* Intravenous bisphosphonate
* Pregnancy
* Smokers, alcoholics and drug abusers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of bone quality | 4 months
  Histomorphometric analysis (Masson's Trichrome stain)

SECONDARY OUTCOMES:
Horizontal ridge dimensional changes | 4 months
  Measuring the linear horizontal changes using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes